

Protocol Number: THR-1442-C-453 Last Revision Date: 07-Apr-2017

# STATISTICAL ANALYSIS PLAN

**Trial Sponsor:** Theracos Sub, LLC. **Protocol Number:** THR-1442-C-453

**IND Number:** 103822

Investigational Drug:Bexagliflozin TabletsIndication:Type 2 Diabetes MellitusDosage Form/Strength:Tablets/20 mg - Bexagliflozin

**Protocol Title:** A Phase 1, Open-label, Randomized, Three-Period, Crossover Study to Evaluate Pharmacokinetic Interaction Between Bexagliflozin Tablets and Metformin, Glimepiride, or Sitagliptin in Healthy Subjects

**Last Revision Date:** 07-Apr-2017

The information contained in this statistical analysis plan is confidential and provided only to Theracos Sub, LLC. Therefore, the information may not be disclosed to, used, or copied by any third party without the written consent of Theracos Sub, LLC or to the extent required by applicable laws, rules and regulations.



Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

# FIRST SIGN-OFF APPROVAL

| Study | Erin Lepic | |
|---|---|---|
| Biostatistician: | Senior Pharmacokinetic Scientist/Project Lead | |
| | Everest Clinical Research | |
| | Lun Lepie | 07-apr-2017 |
| | Signature | 07-Cipe-2017<br>Date |
| Peer Review | Sharon Hunter Senior Biostatistician II Everest Clinical Research Sharon Hunter Sharon Hunter | |
| Biostatistician: | Senior Biostatistician II | |
| | Everest Clinical Research | |
| | Sharen House | 11 1 1 0 1 10 |
| | | 11-1911-6017 |
| | Signature | 11-April - 2017<br>Date |
| Peer Review | Michael Edwardes | |
| Biostatistician: | Principal Biostatistician | |
| | Everest Clinical Research | |
| | OMA A | 7 100 0 7 |
| | - Policeurs | 07-APR-2017 |
| | Signature / | Date |
| Approved by: | Annie Lee Conery | |
| | Clinical Trial Manager | |
| | Translational Medicine Group | |
| | Massachusetts General Hospital | |
| | Strong | 12 - Aρr - 2017 <br> Date |
| | Signature | Date |
| | Xiaoyan Li | |
| | Clinical Trial Manager | |
| | Translational Medicine Group | |
| | Massachusetts General Hospital | |
| | <b>0</b> - | |
| | Signature | 12-APR-2017 |
| | Signature | Date |



Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

# CHANGE LOG FOR CHANGES MADE AFTER THE INITIAL APPROVAL

| Revision | Section(s) | Brief Description of Revision(s) or | Modifications Reviewed and<br>Approved by* |
|---|---|---|---|
| Date** | Modified | Reason(s) for Revision | Sponsor, Everest |

<sup>\*</sup> Provide person's initial and last name.

<sup>\*\*</sup> Update the Last Revision Dates on the cover page and the document header.

Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

# TABLE OF CONTENTS

| 1. | IN | TRODUCTION | 10 |
|----|-----|----------------------------------------------|----|
| 2. | ST | UDY OBJECTIVES | 10 |
| | 2.1 | PRIMARY OBJECTIVE | 10 |
| | 2.2 | SECONDARY OBJECTIVES | 11 |
| 3. | ST | UDY DESIGN | 11 |
| | 3.1 | STUDY DESIGN | 11 |
| | 3.2 | RANDOMIZATION | |
| | 3.3 | Hypothesis Testing | |
| | 3.4 | INTERIM ANALYSIS | 12 |
| | 3.5 | SAMPLE SIZE | |
| | 3.6 | SCHEDULE OF ASSESSMENTS AND STUDY PROCEDURES | 12 |
| 4. | DA | TA AND ANALYTICAL QUALITY ASSURANCE | 17 |
| 5. | AN | ALYSIS POPULATIONS | 17 |
| | 5.1 | SAFETY POPULATION | 17 |
| | 5.2 | PHARMACOKINETIC POPULATION | 17 |
| | 5.3 | PHARMACODYNAMIC POPULATION | 17 |
| 6. | SP | ECIFICATION OF ENDPOINTS AND VARIABLES | 17 |
| | 6.1 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 17 |
| | | 6.1.1 Study Day and Visit Window Definitions | |
| | 6.2 | PHARMACOKINETICS/PHARMACODYNAMICS | |
| | 6.3 | SAFETY | 20 |
| | | 6.3.1 Study Day and Visit Window Definitions | |
| | | 6.3.2 Extent of Exposure to Study Medication | 20 |
| | | 6.3.3 Adverse Events (AEs) | |
| | | 6.3.4 Laboratory Data | |
| | | 6.3.5 Vital Signs | |
| | | 6.3.6 Electrocardiogram | |
| | | 6.3.7 Physical Examination | |
| | | 6.3.8 Pregnancy Test | |
| | | 6.3.9 Concomitant Medications/Treatments | |
| 7. | PH | ARMACOKINETIC/PHARMACODYNAMIC ANALYSES | |
| | 7.1 | GENERAL CONSIDERATIONS | |
| | 7.2 | PHARMACOKINETIC ANALYSES | |
| | 7.3 | PHARMACODYNAMIC ANALYSES | 27 |
| 8. | ST | ATISTICAL ANALYSIS | |
| | 8.1 | GENERAL DATA HANDLING RULES AND DEFINITIONS | |
| | 8.2 | SUBJECT DISPOSITION | |
| | 8.3 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | |
| | 8.4 | SAFETY ANALYSES | |
| | | 8.4.1 Adverse Events | - |
| | | 8.4.2 Laboratory Data | |
| | | 8.4.4 Electrocardiogram (ECG) | |
| | | o.4.4 Diechocatalogiam (DCO) | 30 |



| | 8.4.5 | Physical examinations | 30 |
|---|---|---|---|
| | 8.4.6 | Physical examinations | 30 |
| 9. | ANALYSES | PERFORMED BEFORE DATABASE CLOSURE | 30 |
| 10. | CHANGES | FROM METHODS PLANNED IN THE PROTOCOL | 30 |
| 11. | STATISTIC | AL SOFTWARE | 30 |
| 12. | REFERENC | CES | 30 |
| 13. | APPENDIX | 1 DATA HANDLING RULES | 31 |
| 14. | APPENDIX | 2 SAS CODE FOR STATISTICAL ANALYSES | 32 |
| 15. | | 3 REFERENCE RANGES AND CLINICALLY RELEVANT CHANGES FROM FOR MARKED LABORATORY ABNORMALITIES | 33 |
| 16. | APPENDIX | 4 MOCKUP TABLES, LISTINGS, AND GRAPHS (TLGS) | 34 |



Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

### **GLOSSARY OF ABBREVIATIONS**

| Abbreviation | Term |
|---|---|
| AE | Adverse Event |
| ALB | albumin |
| ALT | alanine aminotransferase |
| ANOVA | analyses of variance |
| AST | aspartate aminotransferase |
| ATC | anatomic therapeutic class |
| AUC | area under the plasma concentration-time curve |
| $\mathrm{AUC}_{\mathrm{extr}}$ | extrapolated area under the plasma concentration-time curve |
| $\mathrm{AUC}_{0\text{-}\infty}$ | area under the plasma concentration-time curve from Time 0 to infinity |
| $\mathrm{AUC}_{0\text{-t}}$ | area under the plasma concentration-time curve from Time 0 to Time t |
| BLOQ | below the limit of quantitation |
| BMI | body mass index |
| BP | blood pressure |
| BUN | blood urea nitrogen |
| Ca | calcium |
| Cl | chloride |
| $C_{last}$ | concentration corresponding to $T_{last}$ |
| CL/F | apparent oral clearance |
| cm | centimeter |
| $C_{\text{max}}$ | maximum observed plasma concentration |
| CRF | case report form |
| CV | coefficient of variation |
| DBP | diastolic blood pressure |
| DDI | drug-drug interaction |
| dL | deciliter |
| DM | data management |



| Abbreviation | Term |
|------------------------|----------------------------------------------|
| ECG | electrocardiogram |
| FDA | Food and Drug Administration |
| FPG | fasting plasma glucose |
| h | hour(s) |
| HBsAg | hepatitis B surface antigen |
| $HCO_3$ | Bicarbonate |
| Hct | hematocrit |
| HCV | hepatitis C virus |
| HDL-C | high density lipoprotein cholesterol |
| Hgb | hemoglobin |
| ICF | informed consent form |
| IRAE | immediately reportable adverse event |
| K | potassium |
| kg | kilogram |
| KR | Kenward-Roger |
| L | liter |
| $\lambda_{\mathrm{z}}$ | terminal elimination phase rate constant |
| LDL-C | low density lipoprotein cholesterol |
| LLN | lower limit of normal |
| LS | least square |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| min | minute |



| Abbreviation | Term |
|---|---|
| mL | milliliter |
| msec | millisecond |
| Na | sodium |
| NCA | non compartmental analysis |
| NTR | not treatment related, includes unrelated |
| OHA | oral hypoglycemic agent |
| OTC | over the counter |
| PCS | potentially clinically significant |
| PD | pharmacodynamic |
| PE | physical examination |
| PK | pharmacokinetic |
| PR | The period that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex (the onset of ventricular depolarization). |
| PT | preferred term |
| QA | quality assurance |
| QC | quality control |
| QRS | The combination of three of the graphical deflections seen on a typical electrocardiogram. |
| QT | Time from electrocardiogram Q wave to the end of the T wave corresponding to the electrical system |
| QTcB | QT corrected using Bazetts formula [QT/(RR <sup>1/2</sup> )] |
| RBC | red blood cell (count) |
| REML | restricted maximum likelihood |
| RR interval | intra-beat interval |
| SAE | serious adverse event |
| SAP | statistical analysis plan |



| Abbreviation | Term |
|---|---|
| SAS | statistical analysis software |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SOC | system organ class |
| SOP | standard operating procedure |
| $T_{\frac{1}{2}}$ | apparent terminal elimination half-life |
| TC | total cholesterol |
| TEAE | treatment emergent adverse event |
| TG | triglycerides |
| $T_{last}$ | time of last measurable (positive) concentration |
| TLF | table, listing, figure |
| $T_{\text{max}}$ | time of maximum observed plasma concentration |
| TR | Treatment related - includes definitely, probably, possibly, and not likely related |
| T-wave | repolarization of the ventricles |
| UGE | urine glucose excretion |
| ULN | upper limit of normal (value) |
| $V_z/F$ | apparent volume of distribution |
| WBC | white blood cell (count) |
| WHO-DD | World Health Organization Drug Dictionary |



Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) outlines the statistical methods for the display, summary and analysis of data collected within the scope of Theracos Sub LLC protocol Ammendment #1 THR-1442-C-453 dated 29-Oct 2016. As with any SAP, the proposed methods and approaches to the data analysis should be deemed as flexible. The analysis of the data should allow changes in the plan to the extent that deviations from the original plan would provide a more reliable and valid analysis of the data. As such, the statistical analysis to a certain degree is iterative since much of the planning is based on assumptions that require verification. The purpose of this plan is to provide general guidelines from which the analysis will proceed. Nevertheless, deviations from these guidelines must be substantiated by a sound statistical rationale.

This SAP should be read in conjunction with the study protocol and the Case Report Forms (CRFs). This version of the SAP has been developed using the final version of the protocol mentioned above and the final version of the annotated CRFs dated 21-NOV-2016.

The SAP details the analysis of the data collected in the study and the presentation of the results of the analyses. The table, listing, and figure (TLF) shells are displayed in a companion document which provides information on the layout of the data displays.

All statistical analyses will be performed using SAS® version 9.4. Adverse events will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA version 19.1 or newer).

This is a phase 1, open-label, randomized, three-period, crossover study to evaluate pharmacokinetic (PK) interaction between bexagliflozin tablets and metformin, glimepiride, or sitagliptin in healthy subjects. A total of 54 healthy subjects will be enrolled and assigned to three groups of eighteen. Each group will participate in one of three open-label, three treatment period, crossover studies:

Group 1: Bexagliflozin/metformin drug-drug interaction (DDI)

Group 2: Bexagliflozin/glimepiride DDI

Group 3 Bexagliflozin/sitagliptin DDI

For each group, every subject will receive a single dose of bexagliflozin, 20 mg, alone, a single dose of an oral hypoglycemic agent (OHA) (1000 mg metformin, 2 mg glimepiride or 100 mg sitagliptin) alone, and the combination of both (bexagliflozin along with OHA) alternatively in a crossover fashion, in three treatment periods separated by a washout period of at least 7 days. Within each group, subjects will be randomized to one of six treatment sequences in an equal ratio.

(See Protocol Sections 3.1 to 3.3 for details).

#### 2. STUDY OBJECTIVES

### 2.1 Primary Objective

To evaluate whether drug-drug interactions following co-administration of bexagliflozin with commonly prescribed OHAs metformin, glimepiride, or sitagliptin result in any change in the PK of bexagliflozin or each of the OHAs.



Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

# 2.2 Secondary Objectives

To evaluate the safety, tolerability, and pharmacodynamics (PD) of bexagliflozin following single dose administration of the drug in combination with commonly prescribed OHAs.

#### 3. STUDY DESIGN

#### 3.1 Study Design

This is a phase 1, open-label, randomized, three-period, crossover study to evaluate PK interaction between bexagliflozin tablets and metformin, glimepiride, or sitagliptin in healthy subjects. Fifty-four (54) eligible healthy subjects will be enrolled and assigned to three groups of eighteen. Each group will participate in one of three open-label, three treatment period, crossover studies:

Group 1: Bexagliflozin/metformin DDI

Group 2: Bexagliflozin/glimepiride DDI

Group 3 Bexagliflozin/sitagliptin DDI

For each group, every subject will receive a single dose of bexagliflozin tablet, 20 mg, alone, a single dose of an OHA (1000 mg metformin, 2 mg glimepiride, or 100 mg sitagliptin) alone, and the combination of both (bexagliflozin tablet and OHA) alternatively in a crossover fashion, in three treatment periods separated by a washout period of at least 7 days. Within each group, subjects will be randomized to one of six treatment sequences in an equal ratio as shown in Table 1 below.

Table 1

| Treatment Sequence | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 |
|---|---|---|---|
| 1 | Bexa alone <sup>1</sup> | OHA alone <sup>2</sup> | Bexa + OHA |
| 2 | Bexa alone | Bexa + OHA | OHA alone |
| 3 | OHA alone | Bexa alone | Bexa + OHA |
| 4 | OHA alone | Bexa + OHA | Bexa alone |
| 5 | Bexa + OHA | OHA alone | Bexa alone |
| 6 | Bexa + OHA | Bexa alone | OHA alone |

<sup>1.</sup> Bexa: bexagliflozin; OHA = oral hypoglycemic agent.

To prevent hypoglycemia, subjects assigned to Group 2 will receive approximately 300 mL of a solution containing 50 g of glucose with study medication at the time of dosing, as well as approximately 75 mL of a solution containing 12.5 g of glucose every 15 minutes for 4 hours post-dose.

During each treatment period for Group 1 (bexagliflozin/metformin DDI) and Group 2 (bexagliflozin/glimepiride DDI), subjects will be admitted to the clinic on the day before dosing and will stay in the clinic until 48 h post-dose. For Group 3 (bexagliflozin/sitagliptin DDI), subjects will stay in the clinic until 72 h post-dose.

For Group 1 and 2, blood samples for PK analysis will be collected in each period prior to dosing (predose) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose. For Group 3, additional PK blood samples will also be collected at 60 and 72 h post-dose.



Protocol No: THR-1442-C-453 Last Revision Date: 07-Apr-2017

Urine samples for PD analysis will be collected in 12 h intervals. For Group 1 and 2, urine samples will be collected pre-dose (-12 to 0 h) and post-dose at 0 to 12 h, 12 to 24 h, 24 to 36 h, and 36 to 48 h. For Group 3, additional samples at 48 to 60 h and 60 to 72 h post-dose will be collected.

Clinical laboratory tests and safety monitoring will be conducted during all treatment periods.

#### 3.2 Randomization

A total of 54 healthy subjects will be enrolled and assigned to one of three groups of eighteen. Each group of eighteen will be randomized to 1 of 6 possible treatment sequences. Subjects who discontinue the study early will not be replaced.

#### 3.3 Hypothesis Testing

No formal statistical hypothesis testing will be conducted for this study.

#### 3.4 Interim Analysis

There will be no interim analysis conducted.

### 3.5 Sample Size

The sample size for this study is not based upon formal statistical consideration. The sample size is considered adequate to characterize the PK of bexagliflozin and OHAs, to assess potential drug-drug interactions, and to provide safety and tolerability data on bexagliflozin when administered alone and in combination with OHAs.

#### 3.6 Schedule of Assessments and Study Procedures



Protocol No. THR-1442-C-453 Last Revision Date: 07-Apr-2017

Table 2. Schedule of Events for Study 1: Bexagliflozin and Metformin Drug-Drug Interaction

| | Screening | | | Perio | 11 | | | | Period 2 | Period 3 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study activity | D -28 to -1 | D0 | D1<br>pre-<br>dose | D1<br>post-<br>dose | D2 | D3 | D7 <sup>1</sup> | D8<br>pre-<br>dose | D8<br>post-<br>dose | D9 | D10 | D14 <sup>1</sup> | D15<br>pre-<br>dose | D15<br>post-<br>dose | D16 | D17 |
| Informed consent form | X | | | | | | | | | | | | | | | |
| Screening for I/E criteria | X | X | | | | | X | | | | | X | | | | |
| Physical examination <sup>2</sup> | X | X | | | | | | | | | | | | | | X |
| Medical history and demographics | X | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | |
| Admission and discharge | | X | | | | X | X | | | | X | X | | | | X |
| Vital signs <sup>3</sup> | X | | X | X | | X | | X | X | | X | | X | X | | X |
| ECG <sup>4</sup> | X | | X | X | | | | X | X | | | | X | X | | X |
| Urinalysis <sup>5</sup> | X | | X | | | X | | X | | | X | | X | | | X |
| Blood draw for clinical lab tests <sup>6</sup> | X | | X | | | X | | X | | | X | | X | | | X |
| Blood sample for PK <sup>7</sup> | | | X | X | X | X | | X | X | X | X | | X | X | X | X |
| Urine Collection for PD <sup>8</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urine Pregnancy Test | X | X | | | | | X | | | | | X | | | | |
| Adverse event and concomitant medication | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study completion | | | | • | | | | • | | | | | | • | • | X |

Abbreviations: D = day; ECG = electrocardiogram; I/E = inclusion/exclusion; PD = pharmacodynamic; PK = pharmacokinetic.

- The admission day for Period 2 and 3 will be 4-6 days after discharge from the previous period.
- 2. A complete physical examination will be performed at screening and day 17 prior to discharge. A partial physical exam will be performed on admission day of Period 1. 3.
- On days 1, 8 and 15, vital signs will be determined at pre-dose and at 4 h and 48 h (day 3, 10 and 17) post-dose.
- ECG data will be recorded at screening, on days 1, 8 and 15 at pre-dose and at 4 h post-dose, at the study termination visit and when clinically indicated.
- Urine samples will be collected for urinalysis at screening, pre-dose and prior to discharge. If urine is dipstick positive for leukocyte esterase or nitrites, sample will be sent for microscopic evaluation and culture. Urine drug screen will only be performed at screening, and if it is conducted more than 5 days prior to dosing, screening shall be repeated.
- Blood samples will be drawn for clinical laboratory tests at screening, pre-dose and prior to discharge. Clinical laboratory tests are listed in Table 2 of the protocol.
- Plasma samples for PK analysis will be collected as described in Section 6.6.2.4 of the protocol.
- Urine collection for the evaluation of urinary glucose and creatinine are described in Section 6.6.2.3 of the protocol.


Table 3. Schedule of Events for Study 2: Bexagliflozin and Glimepiride Drug-Drug Interaction

| | Screening | | | Period 1 | | | | | Period 2 | | Period 3 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study activity | D -28 to -1 | D0 | D1<br>pre-<br>dose | D1<br>post-<br>dose | D2 | D3 | D7 <sup>1</sup> | D8<br>pre-<br>dose | D8<br>post-<br>dose | <b>D9</b> | D10 | D14 <sup>1</sup> | D15<br>pre-<br>dose | D15<br>post-<br>dose | D16 | D17 |
| Informed consent form | X | | | | | | | - | - | - | | | | | | - |
| Screening for I/E criteria | X | X | | | | | X | | | | | X | | | | |
| Physical examination <sup>2</sup> | X | X | | | | | | | | | | | | | | X |
| Medical history and demographics | X | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | |
| Admission and discharge | | X | | | | X | X | | | | X | X | | | | X |
| Vital signs <sup>3</sup> | X | | X | X | | X | | X | X | | X | | X | X | | X |
| ECG <sup>4</sup> | X | | X | X | | | | X | X | | | | X | X | | X |
| Urinalysis <sup>5</sup> | X | | X | | | X | | X | | | X | | X | | | X |
| Blood draw for clinical lab tests <sup>6</sup> | X | | X | | | X | | X | | | X | | X | | | X |
| Blood sample for PK <sup>7</sup> | | | X | X | X | X | | X | X | X | X | | X | X | X | X |
| Urine Collection for PD <sup>8</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urine Pregnancy Test | X | X | | | | | X | | | | | X | | | | |
| Adverse event and concomitant medication | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study completion | | | • | | • | • | | | | | | | | | | X |

Abbreviations: D = day; ECG = electrocardiogram; I/E = inclusion/exclusion; PD = pharmacodynamic; PK = pharmacokinetic.

- The admission day for Period 2 and 3 will be 4-6 days after discharge from the previous period.
- 2. A complete physical examination will be performed at screening and day 17 prior to discharge. A partial physical exam will be performed on admission day of Period 1.
- 3. On days 1, 8 and 15, vital signs will be determined at pre-dose and at 4 h and 48 h (day 3, 10 and 17) post-dose.
- 4. ECG data will be recorded at screening, on days 1, 8 and 15 at pre-dose and at 4 h post-dose, at the study termination visit and when clinically indicated.
- Urine samples will be collected for urinalysis at screening, pre-dose and prior to discharge. If urine is dipstick positive for leukocyte esterase or nitrites, sample will be sent for microscopic evaluation and culture. Urine drug screen will only be performed at screening, and if it is conducted more than 5 days prior to dosing, screening shall be repeated.
- Blood samples will be drawn for clinical laboratory tests at screening, pre-dose and prior to discharge. Clinical laboratory tests are listed in Table 2 of the protocol.
- Plasma samples for PK analysis will be collected as described in Section 6.6.2.4 of the protocol.
- Urine collection for the evaluation of urinary glucose and creatinine are described in Section 6.6.2.3 of the protocol.




Table 4. Schedule of Events for Study 3: Bexagliflozin and Sitagliptin Drug-Drug Interaction

| | Screening | | | Perio | d 1 | | | | | Perio | d 2 | | | Period 3 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study activity | D -28 to<br>-1 | D0 | D1<br>pre-<br>dose | D1<br>post-<br>dose | D2 | D3 | D4 | D7 <sup>1</sup> | D8<br>pre-<br>dose | D8<br>post-<br>dose | D9 | D10 | D11 | <b>D14</b> | D15<br>pre-<br>dose | D15<br>post-<br>dose | D16 | D<br>17 | I<br>1 |
| Informed consent form | X | | | | | | | | | | | | | | | | | | |
| Screening for I/E criteria | X | X | | | | | | X | | | | | | X | | | | | |
| Physical examination <sup>2</sup> | X | X | | | | | | | | | | | | | | | | | 2 |
| Medical history and demographics | X | | | | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | | |
| Admission and discharge | | X | | | | | X | X | | | | | X | X | | | | | Х |
| Vital signs <sup>3</sup> | X | | X | X | | | X | | X | X | | | X | | X | X | | | Х |
| ECG <sup>4</sup> | X | | X | X | | | | | X | X | | | | | X | X | | | Х |
| Urinalysis <sup>5</sup> | X | | X | | | | X | | X | | | | X | | X | | | | Х |
| Blood draw for clinical lab tests <sup>6</sup> | X | | X | | | | X | | X | | | | X | | X | | | | Σ |
| Blood sample for PK <sup>7</sup> | | | X | X | X | X | X | | X | X | X | X | X | | X | X | X | X | Σ |
| Urine Collection for PD <sup>8</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х |
| Urine Pregnancy Test | X | X | | | | | | X | | | | | | X | | | | | |
| Adverse event and concomitant medication | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | 3 |
| Study completion | | | | | • | | | _ | | | | | | | | | | | Σ |

Abbreviations: D = day; ECG = electrocardiogram; I/E = inclusion/exclusion; PD = pharmacodynamic; PK = pharmacokinetic.



- The admission day for Period 2 and 3 will be 3-5 days after discharge from the previous period.
- A complete physical examination will be performed at screening and day 18 prior to discharge. A partial physical exam will be performed on admission day of Period 1.
- On days 1, 8 and 15, vital signs will be determined at pre-dose and at 4 h and 72 h (day 4, 11 and 18) post-dose.
- ECG data will be recorded at screening, on days 1, 8 and 15 at pre-dose and at 4 h post-dose, at the study termination visit and when clinically indicated.
- Urine samples will be collected for urinalysis at screening, pre-dose and prior to discharge. If urine is dipstick positive for leukocyte esterase or nitrites, sample will be sent for microscopic evaluation and culture. Urine drug screen will only be performed at screening, and if it is conducted more than 5 days prior to dosing, screening shall be repeated.
- Blood samples will be drawn for clinical laboratory tests at screening, pre-dose and prior to discharge. Clinical laboratory tests are listed in Table 2 of the protocol.
- Plasma samples for PK analysis will be collected as described in Section 6.6.2.4 of the protocol.
- 8. Urine collection for the evaluation of urinary glucose and creatinine are described in Section 6.6.2.3 of the protocol.




#### 4. DATA AND ANALYTICAL QUALITY ASSURANCE

The overall quality assurance (QA) procedures for the study data, statistical programming and analyses are described in Everest's Standard Operating Procedures (SOPs). Detailed data management (DM) procedures are documented in the Data Management Plan, Data Validation Check Specifications, and Data Review Plan. Detailed statistical and programming quality control (QC) and QA procedures are documented in the Statistical Analysis and Programming QC/QA Plan.

The study endpoints and analytic approaches are both prospectively defined and documented in the protocol and in this SAP. The SAP will be finalized, and protocol violations will be identified and decisions for inclusion and exclusion of subjects from the PK Population will be made prior to the database lock and data analysis.

#### 5. ANALYSIS POPULATIONS

Three subject populations will be evaluated during this study and are defined as follows:

### **5.1 Safety Population**

The Safety Population will include all randomized subjects who receive at least one dose of the investigational product. Subjects will be analyzed according to the treatment received.

### 5.2 Pharmacokinetic Population

The PK Population will include all randomized subjects who receive at least one dose of the investigational product and who have sufficient plasma bexagliflozin and OHA measurements to derive PK parameters following dosing. The PK Population will be used to summarize the PK parameters.

#### 5.3 Pharmacodynamic Population

The PD Population will include all randomized subjects who receive at least one dose of investigational product and will have had at least 2 batches of 12 h urine collection from which to calculate urine glucose excretion (UGE) measurement following dosing. The PD Population will be used to summarize the PD parameters.

#### 6. SPECIFICATION OF ENDPOINTS AND VARIABLES

### 6.1 Demographic and Baseline Characteristics

Demographic variables consist of the following:

- Age in years (continuous) derived as the integer value of (informed consent date date of birth + 1)/365.25
- Sex
- Race
- Ethnicity

Baseline characteristics consist of the following:

- Body mass index (BMI)
- Weight (kg)




- Height (cm)
- Vital signs
  - o systolic blood pressure (SBP, mmHg)
  - o diastolic blood pressure (DBP, mmHg)
  - o oral temperature (°C)
  - o pulse (beats per minute)
  - o respiration rate
- Electrocardiogram (ECG) parameters
  - o RR interval (msec)
  - o PR interval (msec)
  - o QRS duration (msec)
  - o QT interval (msec)
  - o QTcB interval (msec)
- Medical and surgical history
- Clinical laboratory tests
- Prior and concomitant medication
- Physical examination

### 6.1.1 Study Day and Visit Window Definitions

Table 5. Time Windows for Safety Assessments for Group 1 and Group 2

| Time Windows for Safety Assessments | | | |
|---|---|---|---|
| Scheduled Visit Number | Visit (label) | Time Interval (day) | Target Time Point (day) |
| 1 | Screening | -28 to -1 | -28 to -1 |
| 2 | Day 0 | 0 | 0 |
| 3 | Day 1 | 1 | 1 |
| 4 | Day 2 | 2 | 2 |
| 5 | Day 3 | 3-6 | 3 |
| 6 | Day 7 | 7 | 7 |
| 7 | Day 8 | 8 | 8 |
| 8 | Day 9 | 9 | 9 |
| 9 | Day 10 | 10-13 | 10 |
| 10 | Day 14 | 14 | 14 |
| 11 | Day 15 | 15 | 15 |
| 12 | Day 16 | 16 | 16 |
| 13 | Day 17 | 17 | 17 |




Table 6. Time Windows for Safety Assessments for Group 3

| Time Windows for Safety Assessments | | | |
|---|---|---|---|
| Scheduled Visit Number | Visit (label) | Time Interval (day) | Target Time Point (day) |
| 1 | Screening | -28 to -1 | -28 to -1 |
| 2 | Day 0 | 0 | 0 |
| 3 | Day 1 | 1 | 1 |
| 4 | Day 2 | 2 | 2 |
| 5 | Day 3 | 3 | 3 |
| 6 | Day 4 | 4-6 | 4 |
| 7 | Day 7 | 7 | 7 |
| 8 | Day 8 | 8 | 8 |
| 9 | Day 9 | 9 | 9 |
| 10 | Day 10 | 10- | 10 |
| 11 | Day 11 | 11-13 | 11 |
| 12 | Day 14 | 14 | 14 |
| 13 | Day 15 | 15 | 15 |
| 14 | Day 16 | 16 | 16 |
| 15 | Day 17 | 17 | 17 |
| 16 | Day 18 | 18 | 18 |

Data obtained during unscheduled visits will be allocated to the scheduled visit corresponding to the visit window they fall in as specified in Section 6.1.1. Safety data obtained during unscheduled time points will be allocated to the scheduled time point corresponding to the time window in which they fall. Data will be analyzed based on the nominal visits and nominal time points. If the data from the nominal visit or time point is missing, data from unscheduled visits for the same nominal visit or time point will be used. If multiple unscheduled assessments fall in the same visit window or time point, the non-missing assessment closest to target time point will be selected for analysis.

#### 6.2 Pharmacokinetics/Pharmacodynamics

Pharmacokinetic/pharmacodynamic analysis will be performed on the PK and PD Populations respectively Plasma samples will be analyzed for bexagliflozin, metformin, glimepiride, and sitagliptin concentrations using a validated method.

For all groups, blood samples for PK analysis will be collected in each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post dose. For group 3, additional PK blood samples will also be collected at 60 and 72 h post-dose.

Urine samples for PD analysis will be collected in 12 hr intervals.

For all groups, urine collection in 12 h batches will be performed at pre-dose (-12 to 0 h), and post-dose at 0 to 12 h, 12 to 24 h, 24 to 36 h, and 36 to 48 h. For group 3, additional samples at 48 to 60 h and 60 to 72 h post-dose will be collected.




#### 6.3 Safety

Safety analysis will be performed on the Safety Population.

The safety profile of bexagliflozin and OHAs under investigation will be assessed through the recording, reporting, and analyzing of adverse events, clinical evaluations, and laboratory tests.

Safety variables include the following:

- 1. Adverse events
- 2. Clinical laboratory measurements serum chemistry, hematology, and urinalysis
- 3. Urine drug screen
- 4. Vital signs
- 5. ECG
- 6. Physical examination
- 7. Pregnancy test
- 8. Concomitant medications/treatments

#### 6.3.1 Study Day and Visit Window Definitions

Refer to section 6.1.1 for details.

#### **6.3.2** Extent of Exposure to Study Medication

Subjects who gave consent to participate in the study will be randomly assigned to 1 of 3 groups. Subjects in each group will be randomly assigned to receive 1 of 6 treatment regimens in a crossover fashion with 3 treatment periods separated by a washout period of at least 7 days. Refer to Table 1 under Section 3.1. Up to 2 additional washout days will be allowed.

The dosage of bexagliflozin will be 20 mg.

The dosages for the OHAs are equivalent to the highest single tablet dose available for each OHA (1000 mg metformin, 2 mg glimepiride, or 100 mg sitagliptin), and are within recommended daily dose ranges.

# 6.3.3 Adverse Events (AEs)

Adverse events will be collected and coded using version 19.1 (or newer) of MedDRA. Analysis of adverse events will be carried out on the Safety Population. All adverse events will be included in the individual subject data listings. Only treatment emergent adverse events (TEAEs) will be tabulated in summary tables. The incidence of TEAEs will be presented by treatment. If the AE(s) onset date-time or date occurs after the first dose up until right before the second dose, the AE(s) will be assigned to the first treatment. If the AE(s) onset date-time or date occurs after the second dose up until right before the third dose, the AE(s) will be assigned to the second treatment. Any AE(s) that occur after the third dose up until study termination will be assigned to the third treatment.

All adverse events will be assessed by the investigator(s) with respect to severity, relationship to study drug and seriousness.

If an AE becomes serious during the course of the study, the initial AE will be reported with an end date equal to the start date of the serious adverse event (SAE) and outcome 'did not resolve'. The SAE start date will be the date the AE became serious.




### 6.3.3.1 Treatment-Emergent AE (TEAE)

An adverse event is considered treatment-emergent if the date of onset is on or after the date of first dose of study medication, or worsens during the treatment period (intensity/severity grades worsen).

#### 6.3.3.2 Serious Adverse Events (SAE)

AEs will be categorized as serious or non-serious using the definition specified in Section 6.7 of the study protocol.

### 6.3.3.3 Immediately Reportable AE (IRAE)

An IRAE is any serious adverse event or any adverse event that necessitates discontinuation of the study drug.

#### **6.3.3.4** Adverse Events Counting Rules

- 1. A subject with more than one different AE in a particular system organ class (SOC) will be counted only once in the total of subjects experiencing adverse events in that particular SOC.
- 2. A subject having experienced the same event (AE preferred term) more than once during the study will be counted only once in the number of subjects with that event.
- 3. A subject having experienced the same event (AE preferred term) more than once during the study with a different severity or seriousness, it will be counted only once with the worst grade and seriousness respectively.
- 4. A subject having experienced the same event (AE preferred term) more than once during the study with a different causal relationship to the study drug, it will be counted only once by considering the most-related documented degree of relationship.

#### **6.3.3.5 AE** Severity

Adverse events will be graded on a 3-point scale and reported as indicated on the case report form (CRF). The intensity of an adverse experience will be graded as "Mild", "Moderate", and "Severe" using the criteria specified in Section 6.7 of the study protocol.

#### 6.3.3.6 Relationship to the Investigational Medicinal Product

The relationship of an AE to dosing will be assessed as "Definite", "Probable", "Possible", "Not Likely", or Unrelated using the criteria specified in Section 6.7 of the study protocol.

#### 6.3.3.7 AE with Irregular Start/End Dates

Partial dates may be imputed when appropriate. Imputed dates will be used to determine Study Day.

If a partial date is reported for the start of an AE, a complete date will be imputed by the following algorithm:

1. Only the year is reported: If the subject started receiving study medication in the previous year, then January 1 will be used as the starting date of the event. If the subject started receiving study medication in the year reported, then the date of the first dose of study medication will be used as the start of the event.




2. The month and year is reported: If the subject started receiving study medication prior to the month and year reported, then the first day of the month will be used as the starting date of the event. If the subject started receiving study medication during the month and year reported, then the date of the first dose of study medication will be used as the start of the event.

If a partial date is reported for the end of an adverse event and the adverse event is not continuing, a complete date will be imputed by the following algorithm:

- 1. Only the year is reported: If the subject started receiving study drug in the previous year, then the date of final study contact with the subject will be used as the end of the adverse event. If the subject started receiving study medication in the year reported, then the earlier of December 31 or the date of final study contact with the subject will be used as the end of the adverse event.
- 2. The month and year reported: The earlier of the last date of the month or the date of final contact with the subject will be used as the end of the AE.

The above rules are subject to logical sense, for example, imputed start date should be on or prior to imputed end date.

All AEs will be included in the tabulations regardless the completeness of the onset dates.

#### 6.3.4 Laboratory Data

Clinical laboratory tests on hematology, serum chemistry, electrolytes, and lipids and urinalysis will be performed according to the schedule in Section 3.6. Investigators will assess whether there are any clinically significant abnormalities and record the abnormality on medical history or AE forms.

#### **Conversion to the International System of Units**

All laboratory data will be stored in the database with the units in which they are originally reported. Laboratory data in summary tables and subject data listings will be presented in the International System of Units (SI units; Système International d'Unités). Laboratory data not reported in SI units will be converted to SI units before further processing or data analysis.

#### **Abnormal Values**

Based upon laboratory normal ranges, laboratory test results will be categorized according to the normal range as low, normal and high. Subjects with laboratory data outside the normal range will be listed with abnormal values flagged.



**Urine Pregnancy Test** 

# **Statistical Analysis Plan**


# **Table 6 Clinical Laboratory Tests**

| Table 6 Clinical Laboratory Tests | |
|---|---|
| Hematology | |
| Hematocrit (Hct) | Mean corpuscular volume (MCV) |
| Hemoglobin (Hgb) | Platelet count |
| Mean corpuscular hemoglobin (MCH) | Red blood cell (RBC) count |
| Mean corpuscular hemoglobin concentration (MCHC) | White blood cell (WBC) count with differential |
| Serum Chemistry, Electrolytes, and Lipids | |
| Albumin (ALB) | Calcium (Ca) |
| Alanine aminotransferase (ALT) | Magnesium |
| Aspartate aminotransferase (AST) | Phosphorus |
| Blood urea nitrogen (BUN) | Potassium (K) |
| Glucose | Sodium (Na) |
| Total carbon dioxide | Total bilirubin |
| Creatinine | Direct bilirubin |
| Chloride (Cl) | Uric acid |
| Total protein | Low-density lipoprotein cholesterol (LDL-C), calculated |
| Total cholesterol (TC) | |
| High-density lipoprotein cholesterol (HDL-C) | |
| Triglycerides (TG) | |
| Urinalysis | |
| Appearance | Nitrite |
| Bilirubin | pН |
| Color | Protein |
| Glucose | Specific gravity |
| Ketones | Urobilinogen |
| Microscopic examination of sediment | Leukocyte esterase |
| Urine Collection | |
| Glucose | Creatinine |
| Urine Drug Screen | |
| Amphetamines | Opiates |
| Barbiturates | Benzodiazepines |
| Cocaine Metabolites | Cannabinoids |
| Cotinine | |




#### **Infectious Disease Testing**

Hepatitis B Surface Antigen (HbsAg)

Hepatitis C virus (HCV)

#### 6.3.5 Vital Signs

Vital signs include pulse (beats/min), SBP and DBP (mmHg), oral temperature (°C) and respiration rate (breaths/min).

Vital sign changes from baseline will be summarized by treatment and treatment group.

Baseline values are those measured at last evaluation prior to administration of study drug in each treatment period.

Change from baseline to time point t, denoted Change, will be calculated as:

 $Change_t = Value_t - Value_{Baseline}.$ 

### 6.3.6 Electrocardiogram

ECG parameters, including the RR interval (intra-beat interval), PR interval (the period that extends from the beginning of the P wave [the onset of atrial depolarization] until the beginning of the QRS complex [the onset of ventricular depolarization]), QRS duration, and QT interval (the corrected QT interval is the measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle), will be measured according to the study assessment schedule as specified in Section 3.6. Each ECG will be assessed by the Investigator for signs of ischemia, clinically significant hypertrophy, and clinically significant T-wave (repolarization of the ventricles) abnormalities. Baseline ECGs will be defined as the last evaluation performed prior to the administration of study drug in each treatment period.

ECG changes from baseline will be summarized by treatment and treatment group.

Change from baseline to time point t, denoted Change, will be calculated as:

 $Change_t = Value_t - Value_{Baseline}.$ 

#### **6.3.7 Physical Examination**

A complete PE will include measurement of body weight and height (height will be measured only at screening), general assessment of all body systems including the skin, head, eyes, ears, nose, throat, neck, lungs, heart, abdomen, lymph nodes, and extremities.

Physical examination results will be presented in individual subject data listings.

#### **6.3.8 Pregnancy Test**

Only pregnancies considered by the investigator as related to study treatment (e.g., resulting from an interaction between study drug and a contraceptive medication) are considered AEs unto themselves. However, all pregnancies with an estimated conception date during the AE reporting period, must be recorded in the AE section of the eCRF. This applies to both pregnancies in female subjects and in female partners of male subjects.

#### 6.3.9 Concomitant Medications/Treatments

Concomitant medications administered at the time of randomization and during the study will be recorded on the CRF. The medication name, indication, dose, unit, frequency, route of administration, date(s) of




administration and reason for administration will be recorded. This documentation should continue until discharge from the study.

A concomitant medication is any medication the subject enters the trial taking and is expected to continue taking for some portion of the trial, as well as any medication the subject takes during the course of the trial. All prescription and over-the-counter (OTC) medications (non-prescription drugs), including vitamins and herbal supplements, that subjects receive during the trial must be documented on the CRF. This documentation will continue until the subjects are discharged.

Concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD).

All prior and concomitant medication will be presented in individual subject data listings.

For medications with incomplete dates, imputation will be used to convert to a complete date. Imputed dates will be used to determine Study Day.

Partial medication start dates will be imputed as follows:

- 1. Only the year is reported: If the subject started to receive study drug in the year reported, then the date of the first dose of study drug will be used as the starting date of the medication. Otherwise, January 1 will be used as the start of the medication.
- 2. The month and year is reported: If the subject started to receive study drug during the month and year reported, then the date of first dose of study drug will be used as the starting date of the medication. Otherwise, the first day of the month will be used as the start of the medication.

Partial medication end dates will be imputed for non-ongoing medications as follows:

- 1. Only the year is reported: If the subject stopped to receive study drug in the year reported, then the date of the last dose of study drug will be used as the end date of the medication. Otherwise, December 31 will be used as the end of the medication.
- 2. The month and year is reported: If the subject stopped to receive study drug during the month and year reported, then the date of last dose of study drug will be used as the end date of the medication. Otherwise, the last day of the month will be used as the end of the medication.

The above rules are subject to logical sense, for example, imputed start date should be on or prior to imputed end date.

Verbatim terms will be coded and assigned a preferred (PT) term and an ATC (anatomic therapeutic class) term.

#### 7. PHARMACOKINETIC/PHARMACODYNAMIC ANALYSES

#### 7.1 General Considerations

The PK Population will be used for PK analyses. The PD Population will be used for PD analyses.

Statistical and PK analyses will be performed by Everest Clinical Research. Statistical analysis will be performed using Statistical Analysis Software SAS for Windows® (SAS Institute Inc., USA). Non-compartmental analysis (NCA) will be performed using Phoenix® WinNonlin® 6.4 (Certara, USA).




#### 7.2 Pharmacokinetic Analyses

From the plasma concentration-time data, the following PK parameters will be estimated for each subject where feasible.

Table 7. Pharmacokinetic Parameters

| Pharmacokinetic Parameters | |
|---|---|
| $C_{max}$ | Maximum observed plasma concentration |
| $T_{\text{max}}$ | Time of maximum observed plasma concentration |
| $\lambda_{\mathrm{z}}$ | Terminal elimination phase rate constant |
| T <sub>1/2</sub> | Apparent terminal elimination half life |
| CL/F | Apparent oral clearance |
| $V_z/F$ | Apparent volume of distribution |
| $AUC_{0-t}$ | Area under the plasma concentration-time curve from time 0 to time t (time of last quantifiable plasma concentration) |
| AUC <sub>0-∞</sub> | Area under the plasma concentration-time curve from time 0 to infinity |

 $C_{max}$  and  $T_{max}$  will be obtained directly from experimental observations. If multiple maxima occur at equal concentrations, the first temporal value will be taken.

The apparent terminal elimination half-life,  $T_{1/2}$ , where determinable, will be calculated as the natural log of 2 divided by the terminal phase rate constant,  $\lambda_z$ . The number of data points included in the regression will be determined by visual inspection, but a minimum of three data points in the terminal phase, excluding  $C_{max}$ , is required to estimate  $\lambda_z$ . In order for the selection to take place the adjusted  $r^2$  value reported in Phoenix WinNonlin must be > 0.7.

 $AUC_{0-t}$  and  $AUC_{0-\infty}$  will be calculated using the linear trapezoidal linear interpolation method, using actual elapsed time values. If the actual collection time is unknown the nominal collection time may be used for the purposes of PK parameter estimation. For the purpose of calculating AUC, all missing values will be treated as missing in the PK analysis and excluded from analysis except when they occur at pre-dose where they will be set to zero. All values that were below the limit of quantitation (BLOQ) prior to  $T_{max}$  will be set to zero. BLOQ values that occur after  $T_{max}$  will be set to missing. When  $\geq 2$  consecutive plasma concentrations below the limit of quantitation (BLOQ) are encountered after  $T_{max}$ , these and all subsequent values will be excluded from the analysis.

 $AUC_{0-\infty}$  will be calculated as outlined below:

 $AUC_{0-\infty} = AUC_{last} + (C_{last} / \lambda_z)$ , where  $C_{last}$  is the last temporal quantifiable plasma concentration corresponding to  $T_{last}$ .

The proportion of  $AUC_{0-\infty}$  due to extrapolation ( $AUC_{extr}$ ) will be calculated and expressed as a percentage.  $AUC_{0-\infty}$  values will be considered unreliable estimates if the  $AUC_{extr}$  is greater than 20% and will be excluded from summary tables but will be listed.

CL/F will be calculated as Dose/AUC<sub>0-∞</sub>.

 $V_z/F$  will be calculated as Dose/ $(\lambda_z \times AUC_{0-\infty})$ .

 $T_{\frac{1}{2}}$  will be calculated as  $0.693/\lambda_z$ .




Descriptive statistics for the plasma concentrations of measured analytes by Treatment and Timepoint will be provided for each group. Listings of plasma concentrations by Subject Number, Treatment Group, Treatment, Treatment Period, and Timepoint will also be provided.

To assess the effect of the OHAs metformin, glimepiride, and sitagliptin on the PK of bexagliflozin and vice versa, an analyses of variance (ANOVA) using a linear mixed-effects model will be fitted to the natural logarithmic transformation of PK parameters of bexagliflozin ( $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$ ). The linear mixed-effects model will include subject as a random effect, and treatment, period, and sequence as fixed effects. The 90% confidence intervals (CIs) will be constructed for the (bexagliflozin and OHA in combination) to (bexagliflozin alone) or (OHA alone) ratio of the least squares (LS) geometric means of PK parameters ( $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$ ), with 80-125% defined as the lack of interaction boundaries.

The ratios of geometric least squares means and corresponding 90% CI for the treatment comparison will be determined by exponentiating the mean differences between treatments on the logarithm scale. The intrasubject geometric CV%,  $100\%*\sqrt{\exp(residual)-1}$ , where residual = the residual variance component and where exp is the natural exponential function, will be reported.

The appropriateness of the mixed model will be assessed through residual analyses. Any modifications required due to poor fit will be reported and executed.

Descriptive statistics for the PK parameters  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-\infty}$ ,  $AUC_{0-t}$ , CL/F,  $V_z/F$ ,  $\lambda_z$ , and  $T_{1/2}$  will be tabulated by treatment for each group. Means, standard deviations (SD), medians, ranges (minimum; maximum), and geometric means and coefficients of variation (CV) will be presented for all PK parameters with the exception of  $T_{max}$ . Medians and ranges will be presented for  $T_{max}$ .

A listing of derived PK parameters by Subject Number, Treatment Group, and Treatment Period will be provided.

Refer to Appendix 2 for the SAS code.

#### 7.3 Pharmacodynamic Analyses

Urinary glucose excretion will be determined as a PD parameter at baseline and up to 48 hours (Group 1 and Group 2) and up to 72 hours (Group 3). The DDI effect between bexagliflozin and OHAs will be evaluated by comparing the mean cumulative UGE between subjects taking bexagliflozin or OHA alone and bexagliflozin and OHA in combination.

Descriptive statistics of glucose concentrations and UGE will be summarized by Treatment Group, Treatment, and Timepoint.

The quantity of glucose excreted in urine will be determined by multiplying the urine glucose concentration for each time interval by the volume of urine collected for the corresponding collection interval. The total 24-hour, 48-hour, and 72-hour quantity of glucose excreted in urine will be calculated by adding the amounts collected during each interval.

PD data will also be reported in listings.

The effect of an OHA on the cumulative UGE between subjects administered bexagliflozin alone or in combination with an OHA will be compared. The PD parameters, UGE and UGE normalized by urinary creatinine, including UGE<sub>t1-t2</sub>, in 12 hour and 24 hour increments, and total 24-hour, 48-hour, and 72-hour UGE, will be determined. UGE<sub>t1-t2</sub> (mg) will be derived from urine volume ( $V_{t1-t2}$ , mL) x glucose concentration (mg/dL)/100.




#### 8. STATISTICAL ANALYSIS

#### 8.1 General Data Handling Rules and Definitions

All data collected on CRFs will be provided in listings, except data collected only for confirmation of study entry criteria and for study administrative purposes. If any randomized subject is found to be without valid documented informed consent, that subject's data will be excluded from the report, except as necessary to document the error.

All statistical analyses will be conducted using SAS version 9.4 or newer.

Except where specified, all continuous variables will be summarized with descriptive statistics (the number of non-missing values, mean, standard deviation, median, minimum and maximum) and all categorical variables will be summarized with frequency counts and percentages, by treatment and treatment group. Unless otherwise specified, the mean and median will be displayed to 1 more decimal place than the original data, and standard deviation will be displayed to two more decimal places than the original data. All frequencies will be rounded to 1 decimal place.

Missing data will be maintained as missing unless specified otherwise. For variables where missing data is imputed, the analysis dataset will contain one variable with the imputed value and the original variable with missing maintained as missing.

#### 8.2 Subject Disposition

An overall disposition table for all subjects will be presented. This tabulation will include the number of subjects randomized, treated, completed, and those who discontinued early from the study. The number and percentage of randomized subjects who are included in the PK, Safety and PD Populations will also be tabulated.

Subject disposition by treatment and treatment group, and treatment sequence and treatment group, will also be summarized. These tabulations will include the number of subjects dosed, completed, and those who discontinued early from the study along with the corresponding primary reasons for early termination.

Subjects in the Safety Population who prematurely discontinued from the study will be summarized by primary reason for early termination.

All subjects in the Safety Population will be listed.

#### 8.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized by treatment and treatment group, and by treatment sequence and treatment group, for both the Safety and PK Populations and listed.

Descriptive statistics (n, mean, median, standard deviation, minimum, and maximum) will be presented for continuous variables. Frequency distributions (counts and percentages) will be presented for categorical variables.

Medical and surgical history will be summarized and listed. Physical examination, as well as prior and concomitant medications, will also be listed. Prior and concomitant medications will be listed with the drug names and ATC classification codes based on the data collected in the eCRF. The World Health Organization (WHO) Drug Dictionary, version March 2016 or newer, will be used to classify prior and concomitant medications by therapeutic class and drug name.




Abnormalities in the subjects' medical and surgical histories will be coded using version 19.1 (or newer) of MedDRA Medical Dictionary for Regulatory Activities, and summarized and listed.

### 8.4 Safety Analyses

Safety analyses will be performed using the Safety Population, unless otherwise specified.

Safety measurements will include AEs, clinical laboratory tests (i.e. serum chemistry, hematology and urinalysis), ECGs, physical exams and vital signs. All safety data will be summarized by treatment group and treatment. Baseline values for clinical laboratory tests, vital signs and ECGs will be defined as the last evaluation performed prior to administration of study drug.

#### 8.4.1 Adverse Events

All AEs will be coded to system organ class (SOC), and preferred term (PT), using the latest Medical Dictionary for Regulatory Activities coding dictionary (version to be specified in the clinical study report). All reported AEs will be listed, but only TEAEs will be summarized.

The incidence of all TEAEs will be summarized by treatment group and treatment. In the summary tables, subjects may be counted under multiple SOCs and PTs, but for each SOC and PT, subjects are only counted once. If a subject has the same AE on multiple occasions, the highest severity (severe > moderate > mild) or drug relationship (definite > probable > possible > not likely related > unrelated) recorded for the event will be presented. If severity is missing, subjects will be included as missing (for severity). If drug relationship is missing, subjects will be included in related tables (e.g., considered related). Summary tables will be organized by SOC, then PT.

The following summaries will be presented for TEAEs:

- Overall Summary of TEAEs by Treatment Group and Treatment
- Incidence of TEAEs by Treatment Group, Treatment, System Organ Class, and Preferred Term
- Incidence of Treatment Emergent Serious Adverse Events by Treatment Group, Treatment, System Organ Class, and Preferred Term

Subjects who prematurely discontinued due to TEAEs and subjects with serious TEAEs will be listed.

#### 8.4.2 Laboratory Data

Summary tables for laboratory parameters (including hematology, chemistry, and urinalysis) will be summarized for each treatment group and treatment. Summaries for change from baseline for hematology, chemistry, and urinalysis parameters will include descriptive statistics (the number of non-missing values, mean, standard deviation, median, minimum and maximum) for values and change from baseline values for all continuous variables, and frequency counts and percentages for categorical variables, by treatment. Subjects with laboratory data outside the normal range will be listed with abnormal values flagged.

#### 8.4.3 Vital Signs

Summary tables for vital signs data will include descriptive statistics (the number of non-missing values, mean, standard deviation, median, minimum and maximum) for values and change from baseline values by treatment and treatment group.

A listing of vital signs results will be provided for all subjects in the Safety Population.




### 8.4.4 Electrocardiogram (ECG)

ECG parameters (RR interval, PR interval, QRS duration, QT interval, and QTcB interval) will be summarized by changes from baseline values by treatment and treatment group using descriptive statistics. For each parameter, only subjects who had both baseline and a post-baseline assessment will be included in the summary.

A listing of ECG results will be provided for all subjects in the Safety Population.

#### 8.4.5 Physical examinations

Physical examination results will be presented in individual subject data listings.

#### **8.4.6 Pregnancy Test**

Pregnancy test results prior to treatment will be listed.

#### 9. ANALYSES PERFORMED BEFORE DATABASE CLOSURE

No interim analyses are planned for this study.

#### 10. CHANGES FROM METHODS PLANNED IN THE PROTOCOL

Any changes to methods planned in this SAP will be documented in a revision to this statistical plan prior to database lock, or identified in the clinical study report.

#### 11. STATISTICAL SOFTWARE

The statistical software to be used for generation of the tables, listings, and figures is SAS® version 9.4.

#### 12. REFERENCES

Not Applicable.




# 13. APPENDIX 1 DATA HANDLING RULES

| Category | Description | Data Handling Rules |
|---|---|---|
| Demographics | Age at informed consent | Age = integer ([date of informed consent signed - date of birth + 1]/365.25) |
| | | If in date of birth, only day is missing, it is imputed by 15 <sup>th</sup> of the month of birth; both day and month are missing, it is imputed by July 1 <sup>st</sup> of the year of birth. |
| Baseline | | Baseline was defined as the last assessment made before the dose of the investigational product. |
| Vital | Change from | $Change_t = Value_t - Value_{Baseline}$ |
| Signs/ECG/Lab | baseline | |




### 14. APPENDIX 2 SAS CODE FOR STATISTICAL ANALYSES

This section will be completed after examining the existing data and prior to the final signoff of this SAP.

| Test | Table/Figure | SAS Codes for Modeling |
|---|---|---|
| | PK endpoints requiring ANOVA. | Analysis using PROC MIXED in SAS with SEQ, SUBJ, PERIOD, and TRTP identifying SEQUENCE, SUBJECT, PERIOD and TREATMENT variables. "Y" denotes the response measure (log (AUC), log (CMAX)). "KR" denotes Kenward-Roger method. "CL" denotes confidence limits. |
| | | PROC MIXED METHOD=REML; CLASS SUBJ SEQ PERIOD TRTP; MODEL Y = SEQ PERIOD TRTP/ DDFM=KR; RANDOM SUBJ(SEQ); LSMEANS TRTP/ PDIFF CL ALPHA = 0.10; ESTIMATE 'T/R' TREAT -1 1/CL ALPHA = 0.1; RUN; Anti-log transformation to obtain the geometric means. "GEO" denotes geometric and "LS" denotes least square. |
| | | DATA LSMEANS;<br>SET LSMEAN<br>GEOLSMEAN = EXP(ESTIMATE);<br>RUN; |
| | | Anti-log transformation to obtain the ratio of geometric means (point estimate) and 90% confidence interval (CI) – lower and upper bounds. |
| | | DATA DIFFS; SET ESTIMATE; RATIO = EXP(ESTIMATE)*100; LOWER = EXP(LOWER)*100; UPPER = EXP(UPPER) * 100; RUN; |




# 15. APPENDIX 3 REFERENCE RANGES AND CLINICALLY RELEVANT CHANGES FROM BASELINE FOR MARKED LABORATORY ABNORMALITIES

<To be inserted>




# 16. APPENDIX 4 MOCKUP TABLES, LISTINGS, AND GRAPHS (TLGs)

Mockup tables, listings, and graphs are presented in a separate document.